CLINICAL TRIAL: NCT01390012
Title: Oral Versus Intravenous Dexamethasone in Community-Acquired Pneumonia
Brief Title: Oral Versus Intravenous Dexamethasone
Acronym: OVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, E.M.W. van de Garde, PharmD, Dr., St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: OVID
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone oral (Active Comparator)
  Interventions: Drug: Dexamethasone tablet 6 mg
- Dexamethasone intravenous (Active Comparator)
  Interventions: Drug: Dexamethasone injection 4 mg

INTERVENTIONS:
Drug: Dexamethasone tablet 6 mg — Dexamethasone tablet 6 mg
  Arms: Dexamethasone oral
Drug: Dexamethasone injection 4 mg — Dexamethasone injection 4 mg
  Arms: Dexamethasone intravenous

SUMMARY:
The purpose of this study is to assess bioequivalence for dexamethasone administered orally versus intravenously in patients admitted to hospital for pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Presenting to the emergency room with suspected pneumonia (to be confirmed within 24 hours from admission) Pneumonia is defined as a new or progressive infiltrate on a chest X-ray plus at least two of the following criteria: cough, sputum production, temperature >38°C or <35°C, auscultatory findings consistent with pneumonia, leucocytosis or leucopenia (>10 g/l, <4 g/l or >10% rods in leucocyte differentiation), C-reactive protein >3 times the upper normal limit Corticosteroid naive at time of presentation

Exclusion Criteria:

* Patients needing corticosteroid treatment above study medication
* Failure to obtain written consent to participate
* Patients using medication drugs that interact with dexamethasone (i.e. phenytoin, barbiturates, rifampicin, erythromycin, clarithromycin, aprepitant, colchicine, everolimus, itraconazole, ketoconazole, pazopanib, tipranavir, and vinorelbine)
* Moribund patients (defined as expected to die within 24 hours)
* Patients with proven or suspected allergy to dexamethasone
* Patients not capable of taking tablets orally

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration time curve | 0-24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- St. Antonius hospital, Nieuwegein, Utrecht, Netherlands

REFERENCES:
- [Result] Spoorenberg SM, Deneer VH, Grutters JC, Pulles AE, Voorn GP, Rijkers GT, Bos WJ, van de Garde EM. Pharmacokinetics of oral vs. intravenous dexamethasone in patients hospitalized with community-acquired pneumonia. Br J Clin Pharmacol. 2014 Jul;78(1):78-83. doi: 10.1111/bcp.12295. PMID 24400953